CLINICAL TRIAL: NCT06978634
Title: The Effect of SBAR Communication Program on Nursing Students' Perceptions of Clinical Decision Making and Medical Error Prevention Levels: A Mixed Methods Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aytap DİNCER (Other)
Responsible Party: Sponsor-Investigator, Aytap DİNCER, Research Assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B.30.2.ATA.0.01.00/
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Mixed Method Implementation Study; Nursing; Nursing Students; Nursing Education Research
Keywords: SBAR; nursing; nursing students; communication; medical error; clinical decision making
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): In the control group, students who agree to participate in the study and meet the inclusion criteria will receive written permission with a voluntary consent form. The researcher will meet with the students one-on-one and provide information about the purpose of the study. Pre-test data for the study will be collected before the SBAR training with cases. Post-test data will be collected 4 weeks after the training given to the intervention group.
  Students in the control group will receive no intervention and continue with their standard nursing education. They will complete only the pre-test and post-test and will not participate in the SBAR training. Their data will serve as a comparison to evaluate the effectiveness of the intervention.
- intervention (Experimental): The researcher will hold a face-to-face meeting with the students in the intervention group and provide information about the purpose of the study, the content of the training, the Student Guidelines for the SBAR Role Playing Application and the research process. Then, "SBAR Training with Cases" will be given. In addition, a group will be established via Whatsapp and communication during the process will be provided through this channel. The days and times of the training will be determined by looking at the students' course schedules. The training will be carried out in the Skills Laboratory of the Faculty of Health Sciences at Yüzüncü Yıl University.
  Interventions: Other: SBAR training with cases

INTERVENTIONS:
Other: SBAR training with cases — The researcher will hold a face-to-face meeting with the students in the intervention group and provide information about the purpose of the study, the content of the training, the Student Guidelines for the SBAR Role Playing Application and the research process. Then, "SBAR Training with Cases" will be given. In addition, a group will be established via Whatsapp and communication during the process will be provided through this channel. The days and times of the training will be determined by looking at the students' course schedules. The training will be carried out in the Skills Laboratory of the Faculty of Health Sciences at Yüzüncü Yıl University.
  Arms: intervention

SUMMARY:
In clinical settings, teamwork plays a vital role in improving patient care outcomes. Effective and structured communication within the team ensures that a holistic service is provided to patients. However, unclear and inadequate communication between healthcare professionals is a common problem. Such communication problems can be one of the main factors that compromise patient safety and lead to medication errors. Nurses play a key role in this process as they are the healthcare professionals who interact most with patients. Nurses need to not only correctly understand the instructions to be given to the patient, but also to convey information about the patient clearly and accurately to other nurses, doctors and other members of the healthcare team. In this context, opportunities to communicate using a common language and develop these skills form an essential part of the education of nursing students. The use of structured communication tools, especially SBAR, can play an important role in the prevention of medical errors while improving the clinical decision-making skills of future nurses. The SBAR (Situation, Background, Assessment, Recommendation) communication tool is a structured model used to ensure effective communication in healthcare. "The Effect of SBAR Communication Program on Clinical Decision Making and Medical Error Awareness Levels of Nursing Students: A Mixed Method Study" is a mixed method research using experimental and qualitative research designs. The data of the research will be collected with the "Student Information Form", "Clinical Decision Making Scale in Nursing" and "Medical Error Scale for Nursing Students" "Semi-Structured Interview Form". Quantitative data processing and statistical analysis will be done with SPSS (Statistical Package for the Social Sciences) software. Qualitative data analysis will be done using hand coding and content analysis method. As a result, this research will clearly demonstrate the benefits of integrating communication tools such as SBAR into nursing education, contribute to the development of new methods in education and the reduction of medical errors.

DETAILED DESCRIPTION:
The main purpose of handover communication is stated to provide accurate and up-to-date information about patient care, treatment, service use, current status and expected changes in this situation. Ineffective handovers, such as not providing all necessary information, can pose a danger to patients and staff, lead to irrelevant, repetitive and hypothetical information being communicated in the shift report and can cause misuse of resources. The aim of this study, designed as a mixed method, is to develop and implement a role-playing program with scenarios for nursing students using the SBAR communication technique. In addition, it is to examine students' clinical decision-making and medical error awareness as a result of the program. In this direction, when the literature is examined, it is concluded that the role-playing program conducted by Yu and Kang in 2017 using the SBAR technique with nursing students can be used to improve communication skills in nurse-doctor handover and to develop communicative competence in nursing students. In another study examining the experiences and perspectives of nurses who use the SBAR technique to improve patient care, it has been revealed that there are significant improvements in active patient controls and documentation control. It has also been shown that the use of standard protocols and communication tools for bedside handover improves patient care continuity.

A review of the literature on teaching SBAR to nursing students reveals that a variety of teaching methods are used. Methods such as standard patient video recording and feedback, role playing, and computer training have been used to teach communication skills. Several studies have used a combination of didactic and interactive teaching methods (such as role playing) to teach SBAR and have demonstrated positive effects on nurses' communication knowledge, attitudes, and abilities.

Clinical decision making, data analysis, and the application of these skills in a clinical context are important components of the nursing profession. Rapid decision making by nurses shortens treatment time, promotes care, and reduces treatment costs. On the other hand, failure to make timely and appropriate decisions leads to delays in treatment and waste of resources. Therefore, it affects the quality of care. Moreover, in the organizational context, nurses are members of a clinical team. Teamwork requires continuous decision-making. These decisions can affect teamwork and determine the quality of care. When the literature is examined, a study examining the effect of the SBAR communication program on the clinical decision-making levels of nursing students has shown that SBAR-based education can improve nursing students' communication skills and clinical decision-making skills. Similarly, Oh et al. (2021) showed that SBAR-based simulation learning can improve nursing students' clinical judgments and increase confidence in interprofessional communication. Medical errors often occur after breakdowns in handover communications. An analysis of assessment notes conducted by the Joint Commission shows that more than two-thirds of on-call incidents are caused by communication breakdowns, and at least 50% of them occur during handover. To avoid communication breakdown, the SBAR (Situation, Background, Assessment, and Recommendation) technique provides a standardized communication framework for conveying information to healthcare professionals, especially in critical situations that require immediate intervention. Both the Institute for Healthcare Improvement and the Joint Commission recommend the SBAR tool as one of the ways to improve patient and staff safety with its standardized and easy-to-use format for organizing and sharing clinical data among clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Being a student registered in the nursing department,
* Having clinical practice experience (being a 3rd year student),
* Not being a student in an exchange program such as Erasmus,

Exclusion Criteria:

* Coming with a vertical transfer exam
* No clinical practice experience

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Decision Making in Nursing | 5 week
  It was developed by Jenkins (1983) to measure the perceptions of clinical decision-making of nursing students and nurses. Validity and reliability studies in Türkiye were conducted by Durmaz-Edir and Sarıkaya (2015). The scale; Exploring options and ideas (10 items) (1, 3, 6, 7, 16, 22, 27, 30, 32, 37), exploring goals and values (10 items) (2, 9, 10, 14, 21, 31, 33, 35, 38, 40), evaluating consequences (10 items) (13, 17, 18, 23, 25, 26, 28, 29, 34, 39) and searching for information and adopting new information objectively (10 items) (4, 5, 8, 11, 12, 15, 19, 20, 24), 36 items) consists of four subscales and 40 items. The options on a five-point Likert scale are; (1) Never (2) Rarely (3) Sometimes (4) Often (5) Always. The scale's 22 items (1, 3, 5, 7, 8, 9, 10, 11, 14, 16, 17, 18, 20, 26, 27, 28, 29, 33, 35, 36, 37, 38) have positive and 18 items (2, 4, 6, 12, 13, 15, 19, 21, 22, 23, 24, 25, 30, 31, 32, 34, 39, 40) have negative values. The 18 scale items with negative meanings ar

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided